CLINICAL TRIAL: NCT01291628
Title: A Pilot Study- Prevention of Capecitabine Induced Hand and Foot Syndrome
Brief Title: Prevention of Capecitabine Induced Hand and Foot Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, rinat yerushalmi, Medical Oncologist, Rabin Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Socks
Record Dates: First submitted 2011-02-07; First posted 2011-02-08 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Cancer
Keywords: Capecitabine; Hand and foot syndrome; Socks; Copper; Toxicity
MeSH Terms: conditions — Neoplasms; Hand-Foot Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- socks containing copper-oxide fibers (Experimental)
  Interventions: Device: socks containing copper-oxide fibers

INTERVENTIONS:
Device: socks containing copper-oxide fibers — The patients will use a sock which contains copper fibers. The socks are sold in the free market (different Pharma stores) for various purposes such as prevention of diabetic foot. It is a product of Cupron company EPA :84542-2, 84542-3 from April 30 2009.
  Other Names: Cupron company EPA :84542-2, 84542-3 from April 30 2009.

SUMMARY:
Capecitabine is a common anti cancer drug. One of the most common side effects is a syndrome called hand and foot syndrome which comprises of hands and feet redness, swelling, dryness and painful sores. Quite often the drug dose is reduced to suboptimal level due to this side effect. There is no way to prevent or an effective way to treat this side effect. The investigators aim is to investigate whether wearing socks which contain copper fibers may prevent or alleviate the patient symptoms.

DETAILED DESCRIPTION:
Capecitabine is a common anti cancer drug. One of the most common side effects is a syndrome called hand and foot syndrome which comprises of hands and feet redness, swelling, dryness and painful sores. Quite often the drug dose is reduced to suboptimal level due to this side effect. There is no way to prevent or an effective way to treat this side effect. Our aim is to investigate whether wearing socks which contain copper fibers may prevent or alleviate the patient symptoms.

The patients will use socks containing copper-oxide impregnated fibers which are sold in the Pharma stores without physician's prescription.(EPA numbers 8454-2, 8454-3 from April 30 2009).

Drug Toxicity and skin reaction will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stage IV cancer - treated with Capecitabine

Exclusion Criteria:

* Any patient who can not sign an informed consent
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
skin feet toxicity | 1 year
  within the first year from starting Capecitabine use

CONTACTS AND LOCATIONS:
Overall Officials: Rinat Yerushalmi, MD, Principal Investigator — Rabin Medical Center, Affiliated to Tel-Aviv University, Tel-Aviv, Israel; Aaron Sulkes, MD, Principal Investigator — Rabin Medical Center affilated to Tel-Aviv University, Tel-Aviv, Israel
Locations (1):
- Rabin Medical Center, Oncology department, Petah Tikva, Israel

REFERENCES:
- [Background] Hoff PM, Ansari R, Batist G, Cox J, Kocha W, Kuperminc M, Maroun J, Walde D, Weaver C, Harrison E, Burger HU, Osterwalder B, Wong AO, Wong R. Comparison of oral capecitabine versus intravenous fluorouracil plus leucovorin as first-line treatment in 605 patients with metastatic colorectal cancer: results of a randomized phase III study. J Clin Oncol. 2001 Apr 15;19(8):2282-92. doi: 10.1200/JCO.2001.19.8.2282. PMID 11304782
- [Background] Van Cutsem E, Twelves C, Cassidy J, Allman D, Bajetta E, Boyer M, Bugat R, Findlay M, Frings S, Jahn M, McKendrick J, Osterwalder B, Perez-Manga G, Rosso R, Rougier P, Schmiegel WH, Seitz JF, Thompson P, Vieitez JM, Weitzel C, Harper P; Xeloda Colorectal Cancer Study Group. Oral capecitabine compared with intravenous fluorouracil plus leucovorin in patients with metastatic colorectal cancer: results of a large phase III study. J Clin Oncol. 2001 Nov 1;19(21):4097-106. doi: 10.1200/JCO.2001.19.21.4097. PMID 11689577
- [Background] Abushullaih S, Saad ED, Munsell M, Hoff PM. Incidence and severity of hand-foot syndrome in colorectal cancer patients treated with capecitabine: a single-institution experience. Cancer Invest. 2002;20(1):3-10. doi: 10.1081/cnv-120000360. PMID 11853000
- [Background] Cassidy J, Twelves C, Van Cutsem E, Hoff P, Bajetta E, Boyer M, Bugat R, Burger U, Garin A, Graeven U, McKendric J, Maroun J, Marshall J, Osterwalder B, Perez-Manga G, Rosso R, Rougier P, Schilsky RL; Capecitabine Colorectal Cancer Study Group. First-line oral capecitabine therapy in metastatic colorectal cancer: a favorable safety profile compared with intravenous 5-fluorouracil/leucovorin. Ann Oncol. 2002 Apr;13(4):566-75. doi: 10.1093/annonc/mdf089. PMID 12056707
- [Background] Borkow G, Gabbay J. Putting copper into action: copper-impregnated products with potent biocidal activities. FASEB J. 2004 Nov;18(14):1728-30. doi: 10.1096/fj.04-2029fje. Epub 2004 Sep 2. PMID 15345689
- [Background] Ueda K, Morita J, Yamashita K, Komano T. Inactivation of bacteriophage phi X174 by mitomycin C in the presence of sodium hydrosulfite and cupric ions. Chem Biol Interact. 1980 Feb;29(2):145-58. doi: 10.1016/0009-2797(80)90029-0. PMID 6444372
- [Background] Karlstrom AR, Levine RL. Copper inhibits the protease from human immunodeficiency virus 1 by both cysteine-dependent and cysteine-independent mechanisms. Proc Natl Acad Sci U S A. 1991 Jul 1;88(13):5552-6. doi: 10.1073/pnas.88.13.5552. PMID 2062837
- [Background] Kim JH, Cho H, Ryu SE, Choi MU. Effects of metal ions on the activity of protein tyrosine phosphatase VHR: highly potent and reversible oxidative inactivation by Cu2+ ion. Arch Biochem Biophys. 2000 Oct 1;382(1):72-80. doi: 10.1006/abbi.2000.1996. PMID 11051099
- [Background] Cervantes C, Gutierrez-Corona F. Copper resistance mechanisms in bacteria and fungi. FEMS Microbiol Rev. 1994 Jun;14(2):121-37. doi: 10.1111/j.1574-6976.1994.tb00083.x. PMID 8049096
- [Background] Sen CK, Khanna S, Venojarvi M, Trikha P, Ellison EC, Hunt TK, Roy S. Copper-induced vascular endothelial growth factor expression and wound healing. Am J Physiol Heart Circ Physiol. 2002 May;282(5):H1821-7. doi: 10.1152/ajpheart.01015.2001. PMID 11959648